CLINICAL TRIAL: NCT02533687
Title: Comparison of Two Different Bipolar and A Monopolar Energy Sources During Transurethral Resection of Prostate
Brief Title: Comparison of Different Energy Sources During TUR-P
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to unwillingness of surgeons to use monopolar energy & technical problems
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Murat AKAND, Assistant Professor, M.D., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-TURP-BM-01
Record Dates: First submitted 2015-08-23; First posted 2015-08-27 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Benign Prostatic Hypertrophy
Keywords: prostate; transurethral resection; bipolar; monopolar
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bipolar TURP-1 (Active Comparator): Transurethral resection of prostate (TURP) with bipolar resectoscope (Gyrus brand)
  Interventions: Procedure: Bipolar TURP-1
- Bipolar TURP-2 (Active Comparator): TURP with bipolar resectoscope (Olympus brand)
  Interventions: Procedure: Bipolar TURP-2
- Monopolar TURP (Active Comparator): TURP with monopolar resectoscope (Karl Storz brand)
  Interventions: Procedure: Monopolar TURP

INTERVENTIONS:
Procedure: Bipolar TURP-1 — Bipolar transurethral resection of prostate (TURP)
  Arms: Bipolar TURP-1
Procedure: Bipolar TURP-2 — Bipolar TURP
  Arms: Bipolar TURP-2
Procedure: Monopolar TURP — Monopolar TURP
  Arms: Monopolar TURP

SUMMARY:
With this study, it is aimed to compare the operative results and complication rates in transurethral resection of the prostate (TUR-P) performed by resectoscopes with two different bipolar and a monopolar energy sources.

DETAILED DESCRIPTION:
Following data will be collected and evaluated prospectively for the three groups of patients who will undergo TUR-P due to benign prostate hyperplasia (BPH) with one of the resectoscopes using different energy sources:

1. Preoperative data: age, height, weight, body-mass index, concomitant morbidities, use of any drug, history of operation, duration of lower urinary tract symptoms, history of any previous treatment taken for BPH, serum level of prostate specific antigen, prostate volume, maximum and average urine flow rate, postmicturation residual urine volume, hemoglobin level
2. Operative data: duration of operation, volume of resected tissue, observation of obturator reflex (if any), kind and size of the urethral catheter used
3. Postoperative data: time to removal of urethral catheter, hospitalization duration, change in hemoglobin, rate of blood transfusion, any other complications

ELIGIBILITY:
Inclusion Criteria:

* Having an indication due to BPH
* Aged between 40 and 80 years old

Exclusion Criteria:

* Kidney failure due to BPH
* Any kind of coagulopathy or use of anticoagulants in the preoperative period
* History of any previous open or endoscopic prostate surgery

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Uroflowmetry test | Within the first 30 days after surgery.
  Determining the improvement in maximal urine flow (mL/s) and average urine flow (mL/s).

SECONDARY OUTCOMES:
Overall complication rates | Within the first 30 days after surgery.
  Number of patients with any complications related with TURP (including hemorrhage, blood transfusion, urinary tract infections, urethral strictures) classified according to modified Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Akand, MD, Principal Investigator — Selcuk University, School of Medicine, Department of Urology
Locations (1):
- Selcuk University, School of Medicine, Department of Urology, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Background] Komura K, Inamoto T, Takai T, Uchimoto T, Saito K, Tanda N, Minami K, Uehara H, Takahara K, Hirano H, Nomi H, Kiyama S, Watsuji T, Azuma H. Could transurethral resection of the prostate using the TURis system take over conventional monopolar transurethral resection of the prostate? A randomized controlled trial and midterm results. Urology. 2014 Aug;84(2):405-11. doi: 10.1016/j.urology.2014.04.025. Epub 2014 Jun 21. PMID 24958486
- [Background] Nakamura A, Osonoi T, Terauchi Y. Relationship between urinary sodium excretion and pioglitazone-induced edema. J Diabetes Investig. 2010 Oct 19;1(5):208-11. doi: 10.1111/j.2040-1124.2010.00046.x. PMID 24843434
- [Background] Tang Y, Li J, Pu C, Bai Y, Yuan H, Wei Q, Han P. Bipolar transurethral resection versus monopolar transurethral resection for benign prostatic hypertrophy: a systematic review and meta-analysis. J Endourol. 2014 Sep;28(9):1107-14. doi: 10.1089/end.2014.0188. Epub 2014 Jun 5. PMID 24754254